CLINICAL TRIAL: NCT00020774
Title: A Phase IB Clinical Study Of The Farnesyltransferase Inhibitor SCH 66336 And Gemcitabine In Patients With Resectable Primary Liver Neoplasms
Brief Title: SCH 66336 With or Without Gemcitabine Followed by Surgery Compared With Surgery Alone in Treating Patients With Primary Liver Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068712; UCLA-0002038; NCI-G01-1958
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-07

CONDITIONS: Liver Cancer
Keywords: localized resectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Gemcitabine; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: lonafarnib
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of SCH 66336 with or without gemcitabine followed by surgery with that of surgery alone in treating patients who have primary liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the biologic activity and toxicity of neoadjuvant SCH 66336 with or without gemcitabine followed by surgical resection vs surgical resection alone in patients with resectable primary liver cancer.

OUTLINE: This is a randomized, open-label study. Patients are randomized to one of three treatment arms. Arm I: Patients receive neoadjuvant oral SCH 66336 twice daily for 14 days followed by surgical resection. Arm II: Patients receive neoadjuvant oral SCH 66336 twice daily for 14 days and gemcitabine IV over 30 minutes once weekly for 2 weeks followed by surgical resection. Arm III: Patients undergo surgical resection. Patients receive no neoadjuvant therapy prior to resection.

PROJECTED ACCRUAL: Approximately 30 patients (10 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed resectable primary hepatocellular carcinoma or cholangiocarcinoma
* 18 and over
* Karnofsky 70-100%
* Hematopoietic: Absolute neutrophil count greater than 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL Hepatic:
* Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT or SGPT no greater than 5 times ULN
* Albumin at least 2.5 g/dL INR less than 1.3 Renal:
* Creatinine no greater than 1.5 mg/dL
* Cardiovascular: QTc prolongation no greater than 440 msec Other:
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* At least 6 weeks since prior radiotherapy and recovered
* At least 6 weeks since prior surgery and recovered
* At least 6 weeks since prior systemic therapy and recovered

Exclusion Criteria:

* metastatic disease outside of the liver
* pregnant or nursing
* malabsorption or other gastrointestinal (GI) condition that would preclude ability to take oral medication and/or GI absorption (e.g., partial small bowel obstruction)
* non-malignant systemic disease that would preclude study
* active uncontrolled infection No grade II nausea or grade I vomiting despite antiemetic medication
* concurrent immunotherapy Chemotherapy: No other concurrent chemotherapy
* concurrent hormonal therapy including estrogen therapy
* concurrent oral contraceptives or other hormonal methods Concurrent megestrol acetate allowed
* concurrent corticosteroids (except for nausea/vomiting during gemcitabine administration)
* concurrent CYP3A4 inhibitors or inducers including: Azoles (e.g., itraconazole, clotrimazole, fluconazole, or ketoconazole) Macrolide antibiotics (e.g., azithromycin, clarithromycin, or erythromycin) Cyclosporine Grapefruit Antiepileptic medication (e.g., phenytoin, carbamazepine, or phenobarbital) Antibiotics for tuberculosis (e.g., rifampin or isoniazid)
* concurrent HIV protease inhibitors (e.g., amprenavir, ritonavir, or saquinavir mesylate)
* concurrent cisapride
* other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-10; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael G. Amado, MD, Study Chair — Jonsson Comprehensive Cancer Center